CLINICAL TRIAL: NCT01450943
Title: A Comparative Efficacy Study: Treatments of Non-Healing Diabetic Foot Ulcers
Brief Title: VA MERIT: A Comparative Efficacy Study: Treatment of Non-Healing Diabetic
Acronym: DOLCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SURG-005-10S; 11-04-00618 (Other Grant/Funding Number: VA Northern California Health Care System)
Record Dates: First submitted 2011-10-07; First posted 2011-10-13 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Chronic wounds; Chronic ulcers; Oasis; Dermagraft; Adaptic
MeSH Terms: conditions — Diabetic Foot | interventions — Debridement; Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Standard of care (Active Comparator): debridement, irrigation , PRIMARY dressing Adaptic and Iodosorb, SECONDARY dressing gauze and tape
  Interventions: Device: SECONDARY dressing gauze and tape; Procedure: debridement, irrigation
- Dermagraft (Experimental): debridement, irrigation , PRIMARY dressing Dermagraft and Adaptic, SECONDARY dressing gauze and tape
  Interventions: Device: SECONDARY dressing gauze and tape; Procedure: debridement, irrigation; Device: Dermagraft
- Oasis (Experimental): debridement, irrigation , PRIMARY dressing Oasis and Adaptic, SECONDARY dressing gauze and tape
  Interventions: Device: SECONDARY dressing gauze and tape; Procedure: debridement, irrigation; Device: Oasis

INTERVENTIONS:
Device: SECONDARY dressing gauze and tape — SECONDARY dressing gauze and tape
Procedure: debridement, irrigation — debridement, irrigation
Device: Dermagraft — Dermagraft per company protocol
  Arms: Dermagraft
Device: Oasis — Oasis per company protocol
  Arms: Oasis

SUMMARY:
The primary objective of this study is to assess the effectiveness of cellular dermal replacement tissue vs. non-viable extracellular matrix (ECM) for the treatment of non-healing diabetic foot ulcers. Our hypothesis is that these devices are of equal efficacy.

ELIGIBILITY:
Inclusion Criteria:

(Answering NO will exclude patient):

* An Institutional Review Board (IRB) Informed Consent Form signed and dated prior to any study-related activities.
* The area of the study ulcer after debridement is between 1 cm2 and 25 cm2 at Visit 3/Week 0.
* Subjects between 18 and 85 years of age.
* Subject's highest Ankle-Brachial Pressure Index (ABPI) / Ankle-Arm Index (AAI) is greater than or equal to 0.80 and lower than 1.4 (the highest ABPI/AAI value from three measurements within last 6 months shall apply).or a toe-arm index is equal to or higher than 0.6.
* The patient has one or more diabetic ulcers on the target foot with only one ulcer selected as the study (target) ulcer. The target ulcer must be at least 4 cm from a non-target ulcer and in the Investigator's opinion, be unlikely to coalesce with another ulcer within 12 weeks of randomization.
* Subject's study ulcer is full thickness and does not extend to bone, muscle, or tendon.
* Subject's study ulcer has been present at least 4 weeks prior to the initial screening (Visit 1) or 6 weeks at randomization (Visit 3).
* Subject has been diagnosed with Type 1 or Type 2 diabetes and HbA1c is less than 10%.
* Study ulcer has no clinical feature of infection (2 signs of inflammation and elevated bacterial load of the wound).
* For female subjects of childbearing age potential, the subject has a negative pregnancy test and is not lactating for the duration of the study.
* Subject understands the requirements of this study and is willing to comply with all the study requirements.

Exclusion Criteria:

(Answering YES will exclude patient):

* The subject is diagnosed with cancer and is undergoing treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids less than 30 days before enrollment.
* The subject is diagnosed with HIV/AIDS.
* The subject is diagnosed with any bleeding disorders.
* The subject is diagnosed with any connective tissue diseases.
* For female subjects, the subject is pregnant or lactating.
* The subject has a history of illicit drug use within one year of enrollment.
* In the past year, the subject experiences episodes of drinking more than 5 alcoholic beverages in less than two hours and/or drinking alcohol has become a problem in interpersonal relationships, work, driving and/or their behavior in general.
* The subject has any active infected wounds or osteomyelitis (confirmed by bone biopsy, MRI or bone scan).
* Doppler exam within the last 365 days demonstrating reflux greater than 0.5 seconds.
* The subject is diagnosed with active Charcot as described by Saunder's classification system.
* The subject manifests signs of poor nutritional status and/or albumin level < 2.9.
* The subject has been exposed to Dermagraft and/or Oasis in the last 60 days.
* The study ulcer size is less than 0.5 cm2 or greater than 25 cm2.
* The subject has any porcine allergy or cow product allergy.
* The subject's recent (last 30 days) chemistry tests serum creatinine is 2 times above the upper limit of normal and/or LFT's 3 times above the upper limit of normal.
* Between Visit 1/Week -2 and Visit 3/Week 0 (randomization) the study ulcer has decreased in size by more than 40%, or increased in size by more than 50%.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rivkah R. Isseroff, MD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lev-Tov H, Li CS, Dahle S, Isseroff RR. Cellular versus acellular matrix devices in treatment of diabetic foot ulcers: study protocol for a comparative efficacy randomized controlled trial. Trials. 2013 Jan 9;14:8. doi: 10.1186/1745-6215-14-8. PMID 23298410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 subjects enrolled from which 2 study subjects were not randomized into any groups and were terminated from the study; therefore, we only had overall of 118 study subjects.
Groups:
- Standard of Care: Consist of subjects who were randomized to treatment with standard of Care (SOC) which included debridement, irritation, primary dressing, Adaptic, secondary dressing gauze and tape.
- Dermagraft: These are study subject who were randomized to treatment arm with Dermagraft. Dermagraft is a cryopreserved human fibroblast-derived dermal substitute composed of viable newborn foreskin fibroblasts, seeded onto a bio-absorbable polyglactin mesh.
  The treatment included debridement, irrigation, primary dressing and Dermagraft and Adaptic, and secondary dressing with gauze and tape.
  Dermagraft placed per company protocol
- Oasis: These are study subject who were randomized to treatment arm with Oasis. Oasis is a bio-absorbable ECM derived from porcine small intestinal submucosa. the product is processed using proprietary methods to retain its original structure while stored at room temperature.
  The treatment included debridement, irrigation, primary dressing and Oasis and Adaptic, and secondary dressing with gauze and tape.
  Oasis placed per company protocol
Period: Overall Study
Arm/Group | Standard of Care | Dermagraft | Oasis
Started | 28 | 42 | 48
Completed | 26 | 35 | 42
Not Completed | 2 | 7 | 6
Not completed — Screen failure, loss to follow-up | 2 | 7 | 6

BASELINE CHARACTERISTICS:
Population: Veteran subject patient population
Groups:
- Dermagraft: Study subjects who were randomized to treatment arm with Dermagraft. Dermagraft is a cryopreserved human fibroblast-derived dermal substitute composed of viable newborn foreskin fibroblasts, seeded onto a bio-absorbable polyglactin mesh.
  The treatment included debridement, irrigation, primary dressing and Dermagraft and Adaptic, and secondary dressing with gauze and tape.
  Dermagraft placed per company protocol
- Oasis: Study subjects who were randomized to treatment arm with Oasis. Oasis is a bio-absorbable ECM derived from porcine small intestinal submucosa. the product is processed using proprietary methods to retain its original structure while stored at room temperature.
  The treatment included debridement, irrigation, primary dressing and Oasis and Adaptic, and secondary dressing with gauze and tape.
  Oasis placed per company protocol
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Dermagraft | Oasis | Total
Number analyzed (Participants) | 28 | 42 | 48 | 118
Age, Customized [Mean (Standard Deviation); unit: years] | 63.31 (9.09) | 62.83 (9.3) | 61.88 (8.64) | 62.67 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Study subjects information was directly obtained from the individuals and/or patient medical records Population: Northern California veteran patient population
  Participants
    Analyzed participants: Female | 2 | 0 | 1 | 3
    Analyzed participants: Male | 26 | 42 | 47 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Analyzed participants: Hispanic or Latino | 0 | 3 | 4 | 7
  Analyzed participants: Not Hispanic or Latino | 28 | 39 | 44 | 111
  Analyzed participants: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Analyzed participants: American Indian or Alaska Native | 2 | 0 | 6 | 8
  Analyzed participants: Asian | 0 | 0 | 0 | 0
  Analyzed participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Analyzed participants: Black or African American | 2 | 1 | 6 | 9
  Analyzed participants: White | 21 | 37 | 33 | 91
  Analyzed participants: More than one race | 0 | 0 | 0 | 0
  Analyzed participants: Unknown or Not Reported | 3 | 4 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 42 | 48 | 118
BMI [Median (Standard Deviation); unit: kg/m2] | 36.52 (6.59) | 32.44 (5.32) | 36.51 (11.55) | 35.15 (7.83)

OUTCOME MEASURES:

1. Primary Outcome: Wound Closure by Week 15
Description: The primary outcome of interest is defined as the wound healed completely on or before visit 15, regardless of a later recurrence.
Time Frame: 15 weeks
Population: Primary Outcome results consist of data available for the Northern California Veteran patient population participants who completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care: Consist of subjects who were randomized to treatment with standard of Care (SOC) which included debridement, irritation, primary dressing, Adaptic, secondary dressing gauze and tape without any grafts.
Arm/Group | Standard of Care | Dermagraft | Oasis
Number analyzed (Participants) | 26 | 35 | 42
Participants
  Not Healed | 10 | 15 | 9
  Healed completely | 16 | 20 | 33
Statistical Analysis 1: Comparison: Dermagraft vs Oasis; Test type: Superiority; p = 0.0517, Fisher Exact; Odds Ratio (OR) = 2.712595, 95% CI 2-sided [0.9141 to 8.4839]

2. Secondary Outcome: Wound Closure at 20 Weeks
Description: Complete wound closure at study endpoint. The Secondary outcome of interest is defined as the wound healed completely on or before visit 19, regardless of a later recurrence. The number of subjects analyzed at secondary outcome differs from primary outcome due to some subjects not completing the study.
Time Frame: 20 weeks
Population: Primary Outcome results consist of data still available for the Veteran patient population participants who completed the study.
Measure: Number; unit: Wound Closure in weeks
Arm/Group | Standard of Care | Dermagraft | Oasis
Number analyzed (Participants) | 23 | 34 | 39
Wound Closure in weeks
  Not healed | 5 | 9 | 12
  Healed completely | 18 | 25 | 27
Statistical Analysis 1: Comparison: Dermagraft vs Oasis; Test type: Superiority; p = 0.7974, Fisher Exact; Odds Ratio (OR) = 0.812339, 95% CI 2-sided [0.2543 to 2.5224]

3. Secondary Outcome: Cost Effectiveness
Time Frame: 12 weeks
Population: Data not available because the investigators did not asses the cost effectiveness for the study.
Groups:
- Standard of Care: SOC Group:
  debridement, irrigation , PRIMARY dressing and Adaptic, SECONDARY dressing gauze and tape
  SECONDARY dressing gauze and tape: SECONDARY dressing gauze and tape
  debridement, irrigation: debridement, irrigation
- Dermagraft: Dermagraft Group: debridement, irrigation , PRIMARY dressing Dermagraft and Adaptic, SECONDARY dressing gauze and tape
  SECONDARY dressing gauze and tape: SECONDARY dressing gauze and tape
  debridement, irrigation: debridement, irrigation
  Dermagraft: Dermagraft per company protocol
- Oasis: Oasis Group:
  debridement, irrigation , PRIMARY dressing Oasis and Adaptic, SECONDARY dressing gauze and tape
  SECONDARY dressing gauze and tape: SECONDARY dressing gauze and tape
  debridement, irrigation: debridement, irrigation
  Oasis: Oasis per company protocol
Arm/Group | Standard of Care | Dermagraft | Oasis
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Visits 1-2: consent and screen the subject. Obtain medical history, vitals, concomitant medications, and adverse events recorded. Visit 3: If after two weeks, the subject qualifies to continue, the subject is randomized into one of three groups. Visits 4-15: Subjects follow up weekly for study visit which includes wounds undressed, assessed, cleaned and debrided, traced, photographed, and redressed again. Visit 16-19: These are the follow-up visits. There will be 4 visits spread over 16 weeks.
Description: Adverse events were collected through the patient and/or through patient chart review.
Arm/Group | Standard of Care | Dermagraft | Oasis
All-Cause Mortality (participants affected / at risk) | 5/28 | 6/42 | 10/48
Serious Adverse Events (participants affected / at risk) | 6/28 | 15/42 | 16/48
Other Adverse Events (participants affected / at risk) | 3/28 | 4/42 | 2/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=28) | Dermagraft (N=42) | Oasis (N=48)
Non-study related (Infections and infestations) | 6 (6) | 13 (13) | 16 (16) — Cardiac, acute cholecystitis, suicide ideation
Involved study related foot ulcer (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) — Infection that require in patient IV treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=28) | Dermagraft (N=42) | Oasis (N=48)
Non-study related (Cardiac disorders) | 3 (3) | 4 (4) | 2 (2) — Cardiac, Acute cholecystitis, infections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT01450943/Prot_SAP_000.pdf